CLINICAL TRIAL: NCT02885636
Title: Inhaled Beta-adrenergic Agonists to Treat Pulmonary Vascular Disease in Heart Failure With Preserved EF (BEAT HFpEF): A Randomized Controlled Trial
Acronym: BEAT HFpEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Barry Borlaug, Associate Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-005140A; R01HL128526 (NIH); R01HL126638 (NIH); U01HL125205 (NIH); U10HL110262 (NIH)
Record Dates: First submitted 2016-08-24; First posted 2016-08-31 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Congestive Heart Failure; Heart Failure, Left-Sided; Left-Sided Heart Failure
Keywords: Heart Failure with Preserved Ejection Fraction; Pulmonary Hypertension
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Albuterol; Procaterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhaled albuterol (Experimental): 2.5 mg inhaled albuterol through a high efficiency nebulizer -single dose
  Interventions: Drug: Albuterol
- Inhaled saline placebo (Placebo Comparator): Inhaled saline through a high efficiency nebulizer -single dose
  Interventions: Other: Saline placebo

INTERVENTIONS:
Drug: Albuterol — : Experimental: Inhaled albuterol
  2.5 mg inhaled albuterol through a high efficiency nebulizer as a single dose
  Other Names: Proventil, AccuNeb, Proair, Ventolin, and Vospire
  Arms: Inhaled albuterol
Other: Saline placebo — Saline inhaled through a nebulizer as a single dose
  Arms: Inhaled saline placebo

SUMMARY:
The enormous and rapidly growing burden of Heart Failure with Preserved Ejection Fraction (HFpEF) has led to a need to understand the pathogenesis and treatment options for this morbid disease. Recent research from the investigator's group and others have shown that pulmonary hypertension (PH) is highly prevalent in HFpEF, and right ventricular (RV) dysfunction is present in both early and advanced stages of HFpEF.

These abnormalities in the RV and pulmonary vasculature are coupled with limitations in pulmonary vasodilation during exercise. There are no therapies directly targeted at the pulmonary vasculature that have been clearly shown to be effective in HFpEF. A recent study by Mayo Clinic Investigators has demonstrated pulmonary vasodilation with dobutamine (a beta 2 agonist) in HFpEF. As an intravenous therapy, this is not feasible for outpatient use.

In the proposed randomized, placebo-controlled double blinded trial, the investigators seek to evaluate whether the commonly used inhaled bronchodilator albuterol (a beta 2 agonist), administered through a high-efficiency nebulizer device that achieves true alveolar drug delivery, improves pulmonary vascular resistance (PVR) at rest and during exercise in patients with HFpEF as compared to placebo. This has the potential to lead to a simple cost effective intervention to improve symptoms in HFpEF, and potentially be tested in other World Health Organization (WHO) Pulmonary Hypertension groups. PVR is an excellent surrogate marker for pulmonary vasodilation and has been used in previous early trials of PH therapy.

DETAILED DESCRIPTION:
Preliminary studies to support feasibility: Recent research from the investigator's group has shown that right ventricular (RV) dysfunction is present in a third of patients with HFpEF and the presence of pulmonary vascular disease and pulmonary hypertension (PH) is very high (related to both pulmonary venous hypertension as well as pulmonary vascular disease). Both of these have been associated with adverse outcomes and exercise intolerance but no therapy is currently available directly targeted at the pulmonary vasculature in HFpEF.

The investigators recently demonstrated significant improvements in pulmonary vascular function with dobutamine (a β2 agonist) administered acutely in HFpEF. As an intravenous therapy, this is not suitable for chronic outpatient use. Hospitalized patients with heart failure often demonstrate symptomatic improvement with inhaled β2 agonist therapy, even in the absence of pulmonary disease, and animal studies have also shown improved resolution of pulmonary edema with albuterol. In the proposed randomized, double blinded placebo-controlled trial, the investigators seek to evaluate whether the commonly used inhaled bronchodilator albuterol, administered through a high-efficiency nebulizer device, improves pulmonary vascular function in patients with HFpEF-PH as compared to placebo. This has the potential to lead to a simple cost effective intervention to improve symptoms in HFpEF-PH, and potentially be tested in other WHO PH groups.

In the absence of frank signs of congestive heart failure, patients with early HFpEF can only be reliably diagnosed by exercise right heart catheterization, which is routinely performed at Mayo Clinic as part of the evaluation of patients with unexplained dyspnea. The presence of elevated pulmonary capillary wedge pressures (PCWP) at rest (>15 mmHg) or with exercise (>25 mmHg); and elevated mean pulmonary artery pressures at rest (>25 mm Hg) and with exercise (>40 mmHg) has been used to invasively diagnose HFpEF with exercise pulmonary hypertension with a high degree of validity and reliability. Just as exercise stress unmasks abnormalities in left ventricular (LV) diastolic function in early stage HFpEF, the investigators have very recently shown that exercise stress reveals early abnormalities in pulmonary artery vascular function as compared to controls without HF that are not apparent from resting data alone.

Using objective diagnoses of HFpEF and exercise induced PH, the investigators seek to evaluate the hemodynamic changes with exercise in pulmonary vascular resistance, peak cardiac output and subjective dyspnea before and after inhaled albuterol therapy for pulmonary vasodilation.

Study design: This study will be performed in a randomized, double blind placebo-controlled fashion using inhaled albuterol or inhaled saline (prepared by research pharmacy) administered through a novel high-efficiency nebulizer in a 1:1 fashion. Patients will undergo right heart catheterization (RHC) with expired-gas analysis using high Fidelity micromanometer catheters at rest and with exercise, at baseline and following treatment with study drug, using a novel study design that the investigators have previously utilized and reported. Rest and exercise measurements will be repeated after receiving inhaled albuterol or control therapy.

Patients referred to the cardiac catheterization laboratory for invasive exercise stress testing will be prospectively recruited. Standard RHC using high fidelity micromanometers (Millar Instruments) will be performed at rest and during supine exercise with simultaneous expired gas analysis (MedGraphics) as is our current practice. The protocol is rest-20 Watts exercise x 5 minutes, and then graded workload increases in 10-20 Watt increments (3 minute stages) to exhaustion. Hemodynamic, arterial and mixed venous blood gas and expired gas data are acquired at rest, during each exercise stage and at peak exercise. Venous blood samples will be obtained at rest and at peak exercise. Perceived symptoms of dyspnea and fatigue will be quantified using the Borg dyspnea and effort scores at each stage of exercise. Limited echocardiography will be performed by a cardiologist skilled in imaging focused on measures of RV morphology and function.

After the initial exercise study and hemodynamics have returned to baseline, study drug (normal saline placebo or albuterol 2.5 mg) will be inhaled through a high efficiency nebulizer over 5 minutes. After a 10 minute observation period, resting hemodynamic and expired gas data will be acquired exactly as in the initial run. Subjects will then repeat the 20 Watt x 5 minutes exercise phase. Subjects will repeat exercise only at the 20 Watt stage, rather repeating the entire study. This is done to increase the feasibility and shorten the time of the case. The investigators have previously observed that the vast majority (>85%) of the elevation in cardiac filling pressures and reduction in venous oxygen content in people with HFpEF occurs at the low 20 Watt workload, so repeating exercise hemodynamic assessment at this load should be sufficient to detect any clinically meaningful treatment effect from albuterol.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure with Preserved Ejection Fraction (HFpEF)
* Normal left ventricular ejection fraction (≥50%)
* Elevated Left Ventricular filling pressures at cardiac catheterization (defined as resting Pulmonary Capillary Wedge Pressure>15 mmHg and/or ≥25 mmHg during exercise).

Exclusion Criteria:

* Prior albuterol therapy (within previous 48 hours)
* Current long acting inhaled beta agonist use
* Significant hypokalemia (<3meq/L)
* Significant valvular disease (>moderate left-sided regurgitation, >mild stenosis)
* High output heart failure
* Severe pulmonary disease
* Unstable coronary disease
* Constrictive pericarditis
* Restrictive cardiomyopathy
* Hypertrophic cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-09; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Borlaug, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy YNV, Obokata M, Koepp KE, Egbe AC, Wiley B, Borlaug BA. The beta-Adrenergic Agonist Albuterol Improves Pulmonary Vascular Reserve in Heart Failure With Preserved Ejection Fraction. Circ Res. 2019 Jan 18;124(2):306-314. doi: 10.1161/CIRCRESAHA.118.313832. PMID 30582447
- [Derived] Reddy YNV, Obokata M, Wiley B, Koepp KE, Jorgenson CC, Egbe A, Melenovsky V, Carter RE, Borlaug BA. The haemodynamic basis of lung congestion during exercise in heart failure with preserved ejection fraction. Eur Heart J. 2019 Dec 1;40(45):3721-3730. doi: 10.1093/eurheartj/ehz713. PMID 31609443

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhaled Albuterol: 2.5 mg inhaled albuterol through a high efficiency nebulizer -single dose
  Albuterol: : Experimental: Inhaled albuterol
  2.5 mg inhaled albuterol through a high efficiency nebulizer as a single dose
Period: Overall Study
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (8) | 64 (17) | 66 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 9 | 7 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 33.7 (7) | 35.6 (9.2) | 34.6 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in 20 Watt Exercise Pulmonary Vascular Resistance (PVR)
Description: The exercise PVR at 20 Watts after study drug relative to the exercise PVR at 20 Watts in the initial assessment prior to study drug. This measurement is made by subtracting pulmonary capillary wedge pressure from the mean pulmonary arterial pressure and dividing by cardiac output in liters per minute and reported as wood units. A decrease in PVR measured by wood units would be considered a favorable response.
Time Frame: Baseline, 10 minutes after intervention during exercise
Measure: Mean (Standard Deviation); unit: wood units
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
wood units | -0.6 (0.5) | 0.1 (0.7)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.003, ANCOVA

2. Secondary Outcome: Change in Resting Pulmonary Vascular Resistance
Description: The resting PVR after study drug relative to the resting PVR in the initial assessment prior to study drug. This measurement is made by subtracting pulmonary capillary wedge pressure from the mean pulmonary arterial pressure and dividing by cardiac output in liters per minute and reported as wood units.
Time Frame: Baseline, 10 minutes after intervention
Measure: Mean (Standard Deviation); unit: wood units
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
wood units | -0.6 (0.5) | -0.3 (0.8)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.3, t-test, 2 sided

3. Secondary Outcome: Change in Exercise Pulmonary Capillary Wedge Pressure (PCWP)
Description: Pulmonary capillary wedge pressure was measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter. PCWP position was confirmed by appearance on fluoroscopy, characteristic pressure waveforms, and oximetry.
Time Frame: Baseline, 10 minutes after intervention during exercise
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mm Hg | -2 (6) | -3 (3)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.7, t-test, 2 sided

4. Secondary Outcome: Change in Resting Pulmonary Capillary Wedge Pressure (PCWP)
Description: as for outcome 3
Time Frame: Baseline, 10 minutes after intervention
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mm Hg | -2 (2) | -2 (3)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.9, t-test, 2 sided

5. Secondary Outcome: Change in Exercise Pulmonary Artery Compliance
Description: Pulmonary artery compliance was calculated as the ratio of stroke volume/pulmonary artery pulse pressure.
Time Frame: Baseline, 10 minutes after intervention during exercise
Measure: Mean (Standard Deviation); unit: mL/mm Hg
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mL/mm Hg | 1.6 (1.6) | 0.0 (0.7)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.001, t-test, 2 sided

6. Secondary Outcome: Change in Resting Pulmonary Artery Compliance
Description: Pulmonary artery compliance was calculated as the ratio of stroke volume/pulmonary artery pulse pressure.
Time Frame: Baseline, 10 minutes after intervention
Measure: Mean (Standard Deviation); unit: mL/mm Hg
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mL/mm Hg | 1.2 (1.0) | 0.7 (1.0)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.2, t-test, 2 sided

7. Secondary Outcome: Change in Exercise Pulmonary Artery Pressure
Description: Pulmonary artery pressure was measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter.
Time Frame: Baseline, 10 minutes after intervention during exercise
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mm Hg | -8 (4) | -2 (4)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.0002, t-test, 2 sided

8. Secondary Outcome: Change in Resting Pulmonary Artery Pressure
Description: as for outcome 7
Time Frame: Baseline, 10 minutes after intervention
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mm Hg | -5 (3) | -3 (3)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.08, t-test, 2 sided

9. Secondary Outcome: Change in Exercise Right Atrial Pressure (RA)
Description: RA was measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter.
Time Frame: Baseline, 10 minutes after intervention during exercise
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mm Hg | -5 (3) | -1 (2)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.0007, t-test, 2 sided

10. Secondary Outcome: Change in Resting Right Atrial Pressure (RA)
Description: RA was measured using a high-fidelity micromanometer advanced through the lumen of a fluid-filled catheter.
Time Frame: Baseline, 10 minutes after intervention
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mm Hg | -3 (2) | -1 (2)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.03, t-test, 2 sided

11. Secondary Outcome: Change in Exercise Cardiac Output
Description: Cardiac output was calculated using the direct Fick method of breath-by-breath oxygen consumption (V02)/arterial-venous oxygen content difference (AVO2 diff).
Time Frame: Baseline, 10 minutes after intervention during exercise
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
L/min | 2.0 (2.1) | 0.1 (1.0)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.004, t-test, 2 sided

12. Secondary Outcome: Change in Resting Cardiac Output
Description: as for outcome 11
Time Frame: Baseline, 10 minutes after intervention
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
L/min | 0.6 (1.2) | 0.4 (1.2)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.7, t-test, 2 sided

13. Secondary Outcome: Change in Exercise Pulmonary Elastance
Description: Pulmonary elastance was calculated by the ratio of pulmonary artery systolic pressure/stroke volume.
Time Frame: Baseline, 10 minutes after intervention during exercise
Measure: Mean (Standard Deviation); unit: mm Hg/mL
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mm Hg/mL | -0.17 (0.11) | -0.05 (0.11)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.004, t-test, 2 sided

14. Secondary Outcome: Change in Resting Pulmonary Elastance
Description: Pulmonary elastance was calculated by the ratio of pulmonary artery systolic pressure/stroke volume.
Time Frame: Baseline, 10 minutes after intervention
Measure: Mean (Standard Deviation); unit: mm Hg/mL
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
Number analyzed (Participants) | 15 | 15
mm Hg/mL | -0.11 (0.13) | -0.03 (0.13)
Statistical Analysis 1: Comparison: Inhaled Albuterol vs Inhaled Saline Placebo; Test type: Superiority; p = 0.09, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Subjects were monitored in the recovery area for up to two hours after procedure.
Arm/Group | Inhaled Albuterol | Inhaled Saline Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
This was a proof-of-concept study and chronic effects of albuterol were not examined. Further studies testing more clinically meaningful end points are needed to determine whether beta-agonists will improve patient-centric outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02885636/Prot_SAP_000.pdf